CLINICAL TRIAL: NCT05716282
Title: Estimation of Neuromuscular Transmission Recovery After Rocuronium Induced Block - Validation Study of a New Algorithm
Brief Title: Estimation of Neuromuscular Recovery - a Validation Study
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NMB rec_estimation valid
Record Dates: First submitted 2022-12-26; First posted 2023-02-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Neuromuscular Blockade Monitoring
Keywords: Neuromuscular Blocking Agents; Neuromuscular Monitoring; Neuromuscular Nondepolarizing Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMB estimation group: All patients undergoing surgery with a single dose of 0.6 mg/kg rocuronium and quantitative neuromuscular transmission monitoring by TOFScan at the adductor pollicis.
  Interventions: Other: Accuracy of neuromuscular recovery estimation

INTERVENTIONS:
Other: Accuracy of neuromuscular recovery estimation — Accuracy of the estimation of neuromuscular recovery will be measured as:
  * Correct attribution of the patients to the groups slow, intermediate or fast recovery
  * Real speed of recovery falls between 95 confidence interval of the estimated speed of recovery

SUMMARY:
Neuromuscular blocking (NMB) agents are used in the vast majority of surgical interventions. Although pharmacokinetic and pharmacodynamic data are available, there is a large interindividual variability in the time needed for recovery after neuromuscular blocking agents. In a previous study (NTC03550664) a mathematical model in order to estimate for each patient the time needed for full recovery based on the first measurable elements of train-of-four (TOF) recovery was established. After the first 14 TOF measurements, the estimated time to reach a recovery of 90%, expressed as % of recovery per 10 min, is calculated.

In this study, this algorithm will be evaluated on a new cohort of patients in order to measure its accuracy and precision. Patients scheduled for surgery with a single dose of 0.6 mg/kg of rocuronium will be included in this prospective observational study. Neuromuscular transmission will be measured at the adductor pollicis using the TOFScan (IdMed, Marseille, France), a CE approved, commercially available monitor for neuromuscular transmission. TOF ratios will be measured every 30 s and recorded on a PC connected to the TOFScan. According to our algorithm, patients will be classified as slow, intermediate or fast recovery; speed of recovery will be measured as % of recovery per 10 min. A McNemar test will be used to assess the correct classification of patients in each group. Accuracy of the estimated speed of recovery will be assessed by comparing to the 95% confidence interval of our model. If real speed of recovery falls within the 95% confidence interval of the model, the model will be classified as accurate. These measurements will be done at 2 time points: - first estimation available and - after TOF ratio has recovered to 40%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients scheduled for surgery with a single bolus administration of 0.6 mg/kg of rocuronium

Exclusion Criteria:

* patient refusal to participate
* known or suspected allergy to rocuronium
* Body mass index < 20 kg/m2
* Body mass index > 30 kg/m2
* hepatic insufficiency, either clinical or hepatic test abnormalities
* renal insufficiency defined as a clearance < 40 mL/min (calculated by the Modification of diet in renal disease (MDRD) formula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for surgery with a single bolus administartion of 0.6 mg/kg of rocuronium
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of NMB speed of recovery estimation | 6 hours
  A McNemar test will be used to test the attribution of each patient to one of the groups (slow, intermediate or fast recovery)
Precision of NMB speed of recovery estimation | 6 hours
  Speed of recovery estimation (% per 10 min) will be considered precise if it falls within the 95% confidence interval boundaries of the model

CONTACTS AND LOCATIONS:
Locations (1):
- CUB Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs-Buder T, Schreiber JU, Meistelman C. Monitoring neuromuscular block: an update. Anaesthesia. 2009 Mar;64 Suppl 1:82-9. doi: 10.1111/j.1365-2044.2008.05874.x. PMID 19222435
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Ortega R, Brull SJ, Prielipp R, Gutierrez A, De La Cruz R, Conley CM. Monitoring Neuromuscular Function. N Engl J Med. 2018 Jan 25;378(4):e6. doi: 10.1056/NEJMvcm1603741. No abstract available. PMID 29365307